CLINICAL TRIAL: NCT05852431
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Pegozafermin in Subjects With Severe Hypertriglyceridemia (SHTG): The ENTRUST Study
Brief Title: To Evaluate the Efficacy and Safety of Pegozafermin in Subjects With Severe Hypertriglyceridemia
Acronym: ENTRUST
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: 89bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIO89-100-231; 2023-503576-25-00 (EU CTIS Number)
Record Dates: First submitted 2023-05-02; First posted 2023-05-10 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Severe Hypertriglyceridemia
Keywords: SHTG; Hypertriglyceridemia; Metabolic diseases; Hyperlipidemias; Dyslipidemias; Lipid Metabolism Disorders
MeSH Terms: conditions — Hypertriglyceridemia; Metabolic Diseases; Hyperlipidemias; Dyslipidemias; Lipid Metabolism Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pegozafermin - 30mg once a week (Experimental)
  Interventions: Drug: Pegozafermin
- Pegozafermin - 20mg once a week (Experimental)
  Interventions: Drug: Pegozafermin
- Placebo once a week (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pegozafermin — Subcutaneous injection
  Arms: Pegozafermin - 20mg once a week; Pegozafermin - 30mg once a week
Drug: Placebo — Subcutaneous injection
  Arms: Placebo once a week

SUMMARY:
To determine the effect of Pegozafermin on fasting serum triglyceride levels in subjects with Severe Hypertriglyceridemia (TG ≥500 to ≤2000 mg/dL) after 26 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥22 years
* Willing to enter a medication/lifestyle stabilization period during the screening period, which means maintaining those stable medication, eating, and exercise habits for the duration of the study
* Subjects should be on stable background Lipid Modifying Therapy (LMT) to manage ASCVD for a minimum of 4 weeks prior to first qualifying TG

Exclusion Criteria:

* Positive for hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV)
* Uncontrolled or newly diagnosed (≤3 months since diagnosis) Type 2 diabetes mellitus as determined by the Principal Investigator. Subjects must have HbA1c level ≤9.5% at Screening. Medications for glucose management must be stable for at least 4 weeks prior to Screening
* Type 1 diabetes mellitus
* A history of symptomatic gallstone disease, gallstone pancreatitis (unless treated with cholecystectomy), or any other ongoing symptomatic biliary disease
* Acute pancreatitis within 6 months prior to Screening
* Subjects with chronic pancreatitis
* Known or suspected familial chylomicronemia syndrome (FCS) (Type 1 hyperlipoproteinemia)

Other inclusion and exclusion criteria may apply.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline in fasting TG | 26 weeks

SECONDARY OUTCOMES:
Percent change from baseline in non-high-density lipoprotein cholesterol (non-HDL-C) | 26 weeks
Percent change from baseline in high-density lipoprotein cholesterol (HDL-C) | 26 weeks
Percent change from baseline in very low-density lipoprotein cholesterol (VLDL-C) | 26 weeks
Percent change from baseline in total cholesterol (TC) | 26 weeks
Change from baseline in liver fat by magnetic resonance imaging - whole liver proton density fat fraction (MRI-PDFF) | 26 weeks
Percent change from baseline in apolipoprotein B (apo-B) | 26 weeks
Change in HbA1c at Week 26 for those with baseline ≥7.0% | 26 weeks
Percent change from baseline in fasting TG | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Parli, MD, Study Director — 89bio, Inc.
Locations (155):
- United States (72):
  - 89bio Clinical Study Site, Chandler, Arizona
  - 89bio Clinical Study Site, Peoria, Arizona
  - 89Bio Clinical Study Site, Tucson, Arizona
  - 89bio Clinical Study Site, Conway, Arkansas
  - 89bio Clinical Study Site, Jonesboro, Arkansas
  - 89bio Clinical Study Site, Little Rock, Arkansas
  - 89bio Clinical Trial Site, Huntington Park, California
  - 89Bio Clinical Study Site, Long Beach, California
  - 89bio Clinical Study Site, Los Angeles, California
  - 89bio Clinical Trial Site, Northridge, California
  - 89bio Clinical Trial Site, Panorama City, California
  - 89bio Clinical Study Site, Santa Ana, California
  - 89bio Clinical Trial Site, Santa Ana, California
  - 89bio Clinical Study Site, Thousand Oaks, California
  - 89Bio Clinical Study Site, Tustin, California
  - 89bio Clinical Study Site, Wheat Ridge, Colorado
  - 89bio Clinical Trial Site, Wheat Ridge, Colorado
  - 89bio Clinical Study Site, Bridgeport, Connecticut
  - 89Bio Clinical Study Site, Clearwater, Florida
  - 89bio Clinical Study Site, Clearwater, Florida
  - 89bio Clinical Study Site, Hialeah Gardens, Florida
  - 89Bio Clinical Study Site, Homestead, Florida
  - 89Bio Clinical Study Site, Miami Lakes, Florida
  - 89bio Clinical Study Site, Miramar, Florida
  - 89Bio Clinical Study Site, Orlando, Florida
  - 89bio Clinical Study Site, Panama City, Florida
  - 89bio Clinical Trial Site, Port Orange, Florida
  - 89Bio Clinical Study Site, Tampa, Florida
  - 89bio Clinical Study Site, Atlanta, Georgia
  - 89Bio Clinical Study Site, Columbus, Georgia
  - 89Bio Clinical Study Site, Lawrenceville, Georgia
  - 89Bio Clinical Study Site, Chicago, Illinois
  - 89bio Clinical Study Site, West Des Moines, Iowa
  - 89Bio Clinical Study Site, Wichita, Kansas
  - 89Bio Clinical Study Site, Marrero, Louisiana
  - 89bio Clinical Trial Site, Shreveport, Louisiana
  - 89Bio Clinical Study Site, Oxon Hill, Maryland
  - 89bio Clinical Study Site, Flint, Michigan
  - 89bio Clinical Trial Site, Kansas City, Missouri
  - 89bio Clinical Study Site, St Louis, Missouri
  - 89bio Clinical Study Site, Las Vegas, Nevada
  - 89bio Clinical Study Sites, Sparta, New Jersey
  - 89bio Clinical Study Site, East Syracuse, New York
  - 89bio Clinical Trial Site, New Windsor, New York
  - 89bio Clinical Trial Site, New York, New York
  - 89Bio Clinical Study Site, North Massapequa, New York
  - 89bio Clinical Trial Site, Richmond Hill, New York
  - 89bio Clinical Trial Site, Syracuse, New York
  - 89Bio Clinical Study Site, Morganton, North Carolina
  - 89bio Clinical Study Site, Cincinnati, Ohio
  - 89bio Clinical Trial Site, Columbus, Ohio
  - 89bio Clinical Study Site, Middleburg Heights, Ohio
  - 89bio Clinical Study Site, Stow, Ohio
  - 89bio Clinical Study Site, Oklahoma City, Oklahoma
  - 89Bio Clinical Study Site, Eugene, Oregon
  - 89bio Clinical Study Site, Charleston, South Carolina
  - 89Bio Clinical Study Site, Chattanooga, Tennessee
  - 89bio Clinical Trial Site, Clarksville, Tennessee
  - 89bio Clinical Study Site, Tullahoma, Tennessee
  - 89bio Clinical Study Site, Amarillo, Texas
  - 89 Clinical Study Site, Austin, Texas
  - 89bio Clinical Study Site, Dallas, Texas
  - 89bio Clinical Study Site, Graham, Texas
  - 89bio Clinical Study Site, Houston, Texas
  - 89Bio Clinical Study Site, Lampasas, Texas
  - 89bio Clinical Study Site, Mansfield, Texas
  - 89bio Clinical Trial Site, San Antonio, Texas
  - 89bio Clinical Study Site, San Antonio, Texas
  - 89bio Clinical Study Site, Wichita Falls, Texas
  - 89bio Clinical Trial Site, Salt Lake City, Utah
  - 89Bio Clinical Study Site, Burke, Virginia
  - 89bio Clinical Trial Site, Richmond, Virginia
- Argentina (7):
  - 89bio Clinical Study Site, Rosario, Santa Fe Province
  - 89bio Clinical Study Site, Buenos Aires
  - 89bio Clinical Study Site, Córdoba
  - 89bio Clinical Study Site, Mendoza
  - 89bio Clinical Study Site, Rosario
  - 89bio Clinical Study Site, San Miguel de Tucumán
  - 89bio Clinical Study Site, Viedma
- Austria (2):
  - 89bio Clinical Study Site, Graz
  - 89bio Clinical Trial Site, Vienna
- Belgium (4):
  - 89bio Clinical Study Site, Edegem
  - 89bio Clinical Study Site, Ghent
  - 89bio Clinical Study Site, Haine-Saint-Paul
  - 89bio Clinical Study Site, Yvoir
- Bulgaria (9):
  - 89bio Clinical Trial Site, Botevgrad
  - 89bio Clinical Study Site, Dimitrovgrad
  - 89bio Clinical Trial Site, Plovdiv
  - 89bio Clinical Study Site, Sliven
  - 89bio Clinical Trial Site, Sliven
  - 89bio Clinical Trial Site, Sofia
  - 89bio Clinical Study Site, Sofia
  - 89bio Clinical Study Site, Veliko Tarnovo
  - 89bio Clinical Trial Site, Veliko Tarnovo
- Canada (6):
  - 89bio Clinical Study Site, North Vancouver, British Columbia
  - 89bio Clinical Study Site, Brampton, Ontario
  - 89bio Clinical Study Site, Chicoutimi, Quebec
  - 89bio Clinical Study Site, Laval, Quebec
  - 89bio Clinical Study Site, Montreal, Quebec
  - 89bio Clinical Study Site, Québec, Quebec
- Chile (4):
  - 89bio Clinical Study Site, Concepción
  - 89bio Clinical Study Site, Santiago
  - 89bio Clinical Study Site, Valdivia
  - 89bio Clinical Study Site, Viña del Mar
- Czechia (2):
  - 89bio Clinical Study Site, Brno
  - 89bio Clinical Study Site, Prague
- France (3):
  - 89bio Clinical Study Site, Marseille
  - 89bio Clinical Study Site, Paris
  - 89bio Clinical Study Site, Valenciennes
- Georgia (4):
  - 89bio Clinical Study Site, Batumi
  - 89bio Clinical Trial Site, Kutaisi
  - 89bio Clinical Trial Site, Tbilisi
  - 89bio Clinical Study Site, Tbilisi
- Germany (2):
  - 89bio Clinical Study Site, Essen
  - 89bio Clinical Study Site, Leipzig
- Hungary (4):
  - 89bio Clinical Study Site, Baja
  - 89bio Clinical Trial Site, Balatonfüred
  - 89bio Clinical Trial Site, Budapest
  - 89bio Clinical Study Site, Nyíregyháza
- India (7):
  - 89bio Clinical Study Site, Belagāve
  - 89bio Clinical Study Site, Bīkaner
  - 89bio Clinical Study Site, Dehradun
  - 89bio Clinical Study Site, Jaipur
  - 89bio Clinical Study Site, Nagpur
  - 89bio Clinical Study Site, Pimpri-Chinchwad
  - 89bio Clinical Study Site, Varanasi
- Italy (4):
  - 89bio Cllinical Study Site, Genova
  - 89bio Clinical Study Site, Milan
  - 89bio Clinical Study Site, Modena
  - 89bio Clinical Study Site, Reggio Emilia
- Latvia (3):
  - 89bio Clinical Study Site, Daugavpils
  - 89bio Clinical Trial Site, Riga
  - 89bio Clinical Study Site, Zemgale
- Mexico (6):
  - 89bio Clinical Study Site, Monterrey, Nuevo León
  - 89bio Clinical Study Site, Cuernavaca
  - 89bio Clinical Study Site, General Escobedo
  - 89bio Clinical Study Site, Guadalajara
  - 89bio Clinical Study Site, Querétaro City
  - 89bio Clinical Study Site, Tlalpan
- Poland (5):
  - 89bio Clinical Study Site, Bialystok
  - 89bio Clinical Study Site, Krakow
  - 89bio Clinical Study Site, Lodz
  - 89bio Clinical Study Site, Lublin
  - 89bio Clinical Study Site, Warsaw
- 89Bio Clinical Study Site, San Juan, Puerto Rico
- Spain (8):
  - 89bio Clinical Study Site, Barcelona
  - 89bio Clinical Study Site, Cadiz
  - 89bio Clinical Study Site, Córdoba
  - 89bio Clinical Study Site, Granada
  - 89bio Clinical Study Site, Huelva
  - 89bio Clinical Study Site, Madrid
  - 89bio Clinical Study Site, Málaga
  - 89bio Clinical Study Site, Pamplona
- United Kingdom (2):
  - 89bio Clinical Study Site, Cardiff
  - 89bio Clincal Study Site, London

IPD SHARING:
Plan to Share IPD: No